CLINICAL TRIAL: NCT01003119
Title: Developing and Testing a Computer-Based Alcohol Use Disorder Recovery System
Brief Title: Computer-Based Alcohol Use Disorder Recovery System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SE-2009-0484; R01AA017192 (NIH)
Record Dates: First submitted 2009-10-26; First posted 2009-10-28 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Alcohol Dependence
Keywords: Alcohol addiction; Alcohol treatment; Alcohol recovery; Post residential treatment DSM-IV diagnosis of alcohol dependence
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A CHESS (Experimental): Those in the ACHESS arm will also be given a smart-phone with access to the ACHESS system (the intervention) for a full 12 months. The ACHESS intervention includes: 1) the Core CHESS system that has been tested in several diseases, 2) a proactive computer-based relapse prevention system, 3) data transfer from the phone to a computer accessible by the patient's counselor/care manager, and 4) systems for the patient to maintain contact with his/her Care Manager
  Interventions: Behavioral: Addiction CHESS
- Usual Care (No Intervention): Those randomized into the Usual Care group will receive usual medical care.

INTERVENTIONS:
Behavioral: Addiction CHESS — Smartphone with ACHESS application loaded onto the phone.
  Arms: A CHESS

SUMMARY:
The purpose of this grant is to develop and test a proven computer based quality improvement/behavior change e-Health system (CHESS--Comprehensive Health Enhancement Support System) to help prevent relapse in alcohol dependent patients being discharged from residential treatment. The investigators' primary hypothesis is that ACHESS (Addiction CHESS) will improve competence, relatedness and autonomy, which will reduce the days of risky drinking over a 12-month period.

DETAILED DESCRIPTION:
The system to be tested (ACHESS - Addiction CHESS) will be delivered through a new modality (smart-phone rather than PC) to make access more widespread, focus on new patients (alcohol dependent patients leaving residential care), offer optional audio delivery to improve access for those who have literacy challenges and be enhanced with services tailored to relapse prevention. ACHESS will offer: 1) communication with peer support groups and addiction experts; 2) timely monitoring to assess risk of relapse, 3) reminders and alerts to encourage adherence to therapeutic goals; 4) addiction-related educational material and tools tailored to the needs of the particular patient, 5) access to selected Internet based resources and 6) communication with a care manager. Patients randomly assigned to ACHESS will learn to use it prior to discharge from residential care.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be at least 18 years of age
* All subjects must be willing to participate in the study
* All subjects must be willing to identify two people who could provide contact information about their location for the next year
* If randomized into ACHESS, all subjects must agree to allow monitoring of their ACHESS usage, including internet browsing
* All subjects must pass a literacy test

Exclusion Criteria:

* Homelessness
* Psychiatric or medical condition that precludes participation in the study including: subjects with a history of suicidality, significant developmental/cognitive impairments that limit their ability to understand the material or have vision problems will not be included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2009-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
ACHESS + standard care will reduce days of risky drinking over the 12-month follow-up period as measured by three interviews. The time-line follow-back techniques will be used'. | 12 months

SECONDARY OUTCOMES:
ACHESS will reduce proximal outcomes of cravings and negative affect, and produce distal outcomes of increased complete abstinence from alcohol, days of abstinence and reduced negative consequences of substance use. | 12 mos.

CONTACTS AND LOCATIONS:
Overall Officials: David H Gustafson, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - Fayette Companies, Peoria, Illinois
  - CAB Health and Recovery Services, Boston, Massachusetts

REFERENCES:
- [Background] Gustafson DH, Shaw BR, Isham A, Baker T, Boyle MG, Levy M. Explicating an evidence-based, theoretically informed, mobile technology-based system to improve outcomes for people in recovery for alcohol dependence. Subst Use Misuse. 2011;46(1):96-111. doi: 10.3109/10826084.2011.521413. PMID 21190410
- [Result] McTavish FM, Chih MY, Shah D, Gustafson DH. How Patients Recovering From Alcoholism Use a Smartphone Intervention. J Dual Diagn. 2012;8(4):294-304. doi: 10.1080/15504263.2012.723312. Epub 2012 Nov 8. PMID 23316127
- [Result] Gustafson DH, McTavish FM, Chih MY, Atwood AK, Johnson RA, Boyle MG, Levy MS, Driscoll H, Chisholm SM, Dillenburg L, Isham A, Shah D. A smartphone application to support recovery from alcoholism: a randomized clinical trial. JAMA Psychiatry. 2014 May;71(5):566-72. doi: 10.1001/jamapsychiatry.2013.4642. PMID 24671165
- See also: Project Description — http://chess.wisc.edu/chess/projects/AddictionChess.aspx